CLINICAL TRIAL: NCT05612750
Title: Comparative Effectiveness of Online Cognitive Behavioral Therapy vs. An Online Single-Session Pain Relief Skills Class for Chronic Pain - The PROGRESS Study
Brief Title: Comparative Effectiveness of Online 8-session CBT vs. 1-Session Empowered Relief for Chronic Pain - The PROGRESS Study
Acronym: PROGRESS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Beth Darnall, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB-65439
Record Dates: First submitted 2022-08-05; First posted 2022-11-10 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Pain, Chronic; Lupus; Pelvic Pain
Keywords: Young adult; Lupus; Pelvic Pain; Behavioral Health
MeSH Terms: conditions — Chronic Pain; Pelvic Pain | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: A pragmatic clinical trial randomizing to one of two (standard of care) online group behavioral treatments: (1) 8-session cognitive behavioral therapy for chronic pain (pain-CBT); and (2) single-session pain relief skills intervention for chronic pain (Empowered Relief).
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants and research staff will know arm assignment. Co-investigators, project statisticians, and the protocol director at each study site will remain blinded until final assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Lupus Chronic Pain Cohort (Experimental): 150 participants with Lupus and Chronic Pain
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT); Behavioral: Empowered Relief
- Chronic Pelvic Pain (Experimental): 150 participants with Chronic Pelvic Pain
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT); Behavioral: Empowered Relief
- Young Adult (18-23) Chronic Pain (Experimental): 150 participants ages 18-23 with Chronic Pain
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT); Behavioral: Empowered Relief
- PRIME Sample (Experimental): 1200 participants with chronic pain
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT); Behavioral: Empowered Relief

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy (CBT) — A trained psychologist delivers 8 sessions of low-literacy CBT (the LAMP protocol) to groups of patients who were randomized to this treatment arm.
Behavioral: Empowered Relief — A certified instructor delivers 1 session of pain relief skills intervention (Empowered Relief) to groups of patients who were randomized to this treatment arm.

SUMMARY:
The purpose of this study is to conduct a pragmatic clinical trial comparing the effectiveness of: (1) 8-week cognitive behavioral therapy for chronic pain (pain-CBT; sixteen hours total treatment time); and (2) a 1-session pain relief skills intervention for chronic pain (Empowered Relief; two hours total treatment time).

DETAILED DESCRIPTION:
The purpose of this study is to conduct a pragmatic clinical trial comparing the effectiveness: (1) 8-session cognitive behavioral therapy for chronic pain (pain-CBT); and (2) a 1-session pain relief skills intervention for chronic pain (Empowered Relief). The investigators aim to understand for patients which treatment works best.

Online evidence-based behavioral treatment for pain will greatly expand access to patients across the U.S. living with diverse chronic pain conditions. Results from this study will fill several critical gaps in evidence that are preventing patients and physicians from making informed decisions about their pain care.

This study will provide a low-cost, relatively low-risk, widely available and feasible protocol that directly addresses the needs of millions of community-based outpatients and their physicians.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age or older of either sex (and all genders).
2. Chronic pain (pain that occurs on at least half of the days of 3 months or more).
3. Past-month average pain intensity score of at least 3/10.
4. Ability to adhere to and complete study protocols.

Exclusion Criteria:

1. Inability to provide informed consent.
2. Cognitive impairment, non-English speaking, or psychological factors that would preclude comprehension of material and/or full participation in the study including group treatment.
3. Active suicidality at screening.
4. Study staff may exclude individuals with a known history of disruptive behavior to minimize contamination of the learning environment for an entire treatment cohort.
5. Receipt of either study treatment in the past 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1650 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2029-05-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | 1 months
  Compare study treatments for primary outcomes post-treatment with the Numeric Rating Scale (0-10)
Pain Intensity | 2 months
  Compare study treatments for primary outcomes post-treatment with the Numeric Rating Scale (0-10)
Pain Intensity | 3 months
  Compare study treatments for primary outcomes post-treatment with the Numeric Rating Scale (0-10)
Pain Intensity | 6 months
  Compare study treatments for primary outcomes post-treatment with the Numeric Rating Scale (0-10)
Pain Interference | 1 month
  Compare study treatments for primary outcomes post-treatment with the Numeric Rating Scale (0-10)
Pain Interference | 2 months
  Compare study treatments for primary outcomes post-treatment with the PROMIS Pain Interference 6-item scale.
Pain Interference | 3 months
  Compare study treatments for primary outcomes post-treatment with the PROMIS Pain Interference 6-item scale.
Pain Interference | 6 months
  Compare study treatments for primary outcomes post-treatment with the PROMIS Pain Interference 6-item scale.

SECONDARY OUTCOMES:
Sleep Disturbance | 1 month
  Compare treatment groups on the PROMIS Sleep Disturbance 6-item
Sleep Disturbance | 2 months
  Compare treatment groups on the PROMIS Sleep Disturbance 6-item
Sleep Disturbance | 3 months
  Compare treatment groups on the PROMIS Sleep Disturbance 6-item
Sleep Disturbance | 6 months
  Compare treatment groups on the PROMIS Sleep Disturbance 6-item
Pain Bothersomeness | 1 month
  Compare treatment groups for Pain Bothersomeness on a Numeric Rating Scale (0-10)
Pain Bothersomeness | 2 months
  Compare treatment groups for Pain Bothersomeness on a Numeric Rating Scale (0-10)
Pain Bothersomeness | 3 months
  Compare treatment groups for Pain Bothersomeness on a Numeric Rating Scale (0-10)
Pain Bothersomeness | 6 months
  Compare treatment groups for Pain Bothersomeness on a Numeric Rating Scale (0-10)
Pain Catastrophizing | 1 months
  Pain Catastrophizing Scale is a 13-item measure with a total score ranging from 0-52 with higher scores indicative of more catastrophizing.
Pain Catastrophizing | 2 months
  Pain Catastrophizing Scale is a 13-item measure with a total score ranging from 0-52 with higher scores indicative of more catastrophizing.
Pain Catastrophizing | 3 months
  Pain Catastrophizing Scale is a 13-item measure with a total score ranging from 0-52 with higher scores indicative of more catastrophizing. We aim to obtain >30% reduction in PCS scores after the intervention
Pain Catastrophizing | 6 months
  Pain Catastrophizing Scale is a 13-item measure with a total score ranging from 0-52 with higher scores indicative of more catastrophizing.
Anxiety | 1 month
  Compare treatment groups for anxiety using the PROMIS Anxiety 6-item
Anxiety | 2 months
  Compare treatment groups for anxiety using the PROMIS Anxiety 6-item
Anxiety | 3 months
  Compare treatment groups for anxiety using the PROMIS Anxiety 6-item
Anxiety | 6 months
  Compare treatment groups for anxiety using the PROMIS Anxiety 6-item
Satisfaction with Social Roles/Responsibilities | 1 month
  Compare treatment groups for PROMIS 6 item Satisfaction with Social Roles/Responsibilities
Satisfaction with Social Roles/Responsibilities | 2 months
  Compare treatment groups for PROMIS 6 item Satisfaction with Social Roles/Responsibilities
Satisfaction with Social Roles/Responsibilities | 3 months
  Compare treatment groups for PROMIS 6 item Satisfaction with Social Roles/Responsibilities
Satisfaction with Social Roles/Responsibilities | 6 months
  Compare treatment groups for PROMIS 6 item Satisfaction with Social Roles/Responsibilities
Patient Global Impression of Change | 1months
  Compare treatment groups for PROMISE 1 item Global Impression of Change scale
Patient Global Impression of Change | 2 month
  Compare treatment groups for PROMISE 1 item Global Impression of Change scale
Patient Global Impression of Change | 3 months
  Compare treatment groups for PROMISE 1 item Global Impression of Change scale
Patient Global Impression of Change | 6 months
  Compare treatment groups for PROMISE 1 item Global Impression of Change scale
Depression | 1 month
  Compare study treatments for primary outcomes post-treatment with the PROMIS 6 item Depression scale.
Depression | 2 months
  Compare study treatments for primary outcomes post-treatment with the PROMIS 6 item Depression scale.
Depression | 3 months
  Compare study treatments for primary outcomes post-treatment with the PROMIS 6 item Depression scale.
Depression | 6 months
  Compare study treatments for primary outcomes post-treatment with the PROMIS 6 item Depression scale.
Fatigue | 1 month
  Compare study treatments for primary outcomes post-treatment with the PROMIS 6 item Fatigue scale.
Fatigue | 2 months
  Compare study treatments for primary outcomes post-treatment with the PROMIS 6 item Fatigue scale.
Fatigue | 3 months
  Compare study treatments for primary outcomes post-treatment with the PROMIS 6 item Fatigue scale.
Fatigue | 6 months
  Compare study treatments for primary outcomes post-treatment with the PROMIS 6 item Fatigue scale.
Anger | 1 month
  Compare study treatments for primary outcomes post-treatment with the PROMIS 5 item Anger scale.
Anger | 2 months
  Compare study treatments for primary outcomes post-treatment with the PROMIS 5 item Anger scale.
Anger | 3 months
  Compare study treatments for primary outcomes post-treatment with the PROMIS 5 item Anger scale.
Anger | 6 months
  Compare study treatments for primary outcomes post-treatment with the PROMIS 5 item Anger scale.

OTHER OUTCOMES:
Exploratory Outcome Health Service Utilization | 6 months
  We will utilize EMR and database records to compare treatment groups for healthcare utilization (e.g., medical visits) during final 3 months of the study vs. 3 months prior to enrollment.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Phoenix VA Health Care System, Phoenix, Arizona
  - SCAN Health Plan, Long Beach, California
  - Humana, Louisville, Kentucky
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Intermountain Healthcare, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No